CLINICAL TRIAL: NCT01583855
Title: Manual vs Amigo SmartTouch Atrial Fibrillation Study
Acronym: MAST-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0260
Record Dates: First submitted 2012-02-27; First posted 2012-04-24 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
Keywords: Remote catheter ablation; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual ablation (Active Comparator): Patients will have their ablation performed manually.
  Interventions: Procedure: Catheter ablation for atrial fibrillation, manual
- Ablation using remote catheter system (Active Comparator): Ablation for atrial fibrillation using the Amigo remote catheter system
  Interventions: Device: Ablation using Amigo remote catheter system

INTERVENTIONS:
Procedure: Catheter ablation for atrial fibrillation, manual — Ablation for atrial fibrillation will be performed manually
  Arms: Manual ablation
Device: Ablation using Amigo remote catheter system — Atrial fibrillation ablation will be performed using the Amigo remote catheter system
  Arms: Ablation using remote catheter system

SUMMARY:
Atrial fibrillation is a common form of heart rhythm disturbance that for some patients is treated by catheter ablation (making an ablation lesion or burn inside the heart using a fine wire (catheter)). A new system for manipulating the catheters has recently been introduced into clinical practice (the Amigo Remote Catheter System (RCS)). This trial is designed to answer two primary questions: a) is the contact force (the force with which the catheter comes into contact with the heart) any different using the RCS to manual techniques,and b)are the resulting ablation lesions within the heart any different in terms of the volume and contiguity of the lesions produced. Additionally the investigators aim to determine how the two techniques compare in success (the proportion of patients whose heart rhythm disturbance is corrected by the procedure).

DETAILED DESCRIPTION:
The trial aims to recruit 50 patients, randomised into two groups, to have ablation for atrial fibrillation performed either using the RCS, or manually. Contact force information will be collected during the procedure, but the operators will be blinded to this information. Patients will have follow-up to include post-procedural cardiac magnetic resonance imaging and ambulatory electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation
* scheduled for catheter ablation

Exclusion Criteria:

* contraindication to magnetic resonance imaging
* pregnancy
* life expectancy of less than six months
* participation in another trial that would conflict with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03-01; Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
Contact force delivered | Contact force information collected at the time of the procedures
  The contact force delivered by the catheter is measured and will be compared between the two groups.

SECONDARY OUTCOMES:
Quantity and contiguity of ablation lesions | 3 months post procedure
  Cardiac magnetic resonance will be used to quantify and assess contiguity of ablation lesions.
Recurrence of atrial fibrillation | 1 year
  Patients will be asked to attend office follow-up up to one year post procedure to assess for recurrence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: G Andre Ng, MBChB, PhD, Principal Investigator — University of Leicester, UK
Locations (1):
- Glenfield Hospital, Groby Road, Leicester, United Kingdom